CLINICAL TRIAL: NCT01108068
Title: Trial of Lithium Carbonate for Treatment of Osteoporosis Pseudoglioma Syndrome
Brief Title: Trial of Lithium Carbonate for Treatment of Osteoporosis-pseudoglioma Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Elizabeth Streeten, Clinical Professor of Medicine, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00040536
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2018-04

CONDITIONS: Osteoporosis Pseudoglioma
Keywords: Osteoporosis-pseudoglioma syndrome, OPPG, LRP5 mutation
MeSH Terms: conditions — Exudative Vitreoretinopathy 4; Osteoporosis-pseudoglioma syndrome | interventions — Lithium; Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lithium (Experimental): patients with OPPG will be treated with lithium for 6 months
  Interventions: Drug: Lithium
- Unaffected controls (No Intervention): Family members of patients with OPPG will have DXA and pQCT to compare to OPPG patients. These unaffected participants will not receive lithium.

INTERVENTIONS:
Drug: Lithium — lithium will be given for 6 months to patients with OPPG, starting at a low dose of 2.5 mg/kg daily, gradually increasing until a lithium blood level of 0.3-0.6 ng/dl is achieved.
  Other Names: lithium carbonate or lithium citrate will be used
  Arms: Lithium

SUMMARY:
This was a pilot study of 10 patients with Osteoporosis-pseudoglioma syndrome (OPPG) from the Old Order Mennonite community and 16 controls, who did not have OPPG. Five of the 10 OPPG patient elected to participate in the Lithium trial and 5 participated only in baseline data (labs, pQCT). The 5 with OPPG who were given lithium for 6 months had both dual energy xray absorptiometry (DXA), peripheral quantitative computerized tomography (pQCT) and lab assessment at baseline and 6 months. Studies in the mouse model of OPPG showed that lithium normalized their bone strength. Controls (n=16) were recruited from the Old Order Mennonite community, to minimize the effects of environmental and lifestyle factors. The controls were not be given lithium. The age range of participants was 4-64 years.

DETAILED DESCRIPTION:
Osteoporosis-pseudoglioma (OPPG) syndrome is a very rare genetic disorder (approximately 50 cases have been reported worldwide) due to mutations in the LRP5 gene, causing blindness from birth and fragile bones (osteoporosis)in early childhood. The bony fragility can lead to recurrent fractures of major bones such as the hip (femur) and spine, leaving some children in wheelchairs.

Treatment to strengthen the bones in OPPG has primarily been with osteoporosis medications used in other fragile bone disorders of childhood and in adults, namely the bisphosphonates (eg. pamidronate, alendronate). These drugs have helped the bone strength in OPPG somewhat but have not prevented all fractures. We have observed fractures of the hip in 3 children with OPPG who we have treated, in spite of their attaining normal bone density (determined by DXA, dual xray absorptiometry) with bisphosphonates. Therefore, new treatments for OPPG are greatly needed and new methods besides DXA are needed to monitor bone strength on treatment.

A mouse model of OPPG has been created. In the mouse model of OPPG, lithium dramatically improved their bones, returning them to normal strength and preventing fractures. Lithium, which is used for people with psychiatric disease, is known to lead to higher bone strength and reduced fractures in people who are on it for psychiatric disease. Lithium has been used safely and is approved for children 12 and above. The theory is that lithium will improve bone strength in OPPG in humans, as it has in the mouse, by stimulating bone production bypassing the genetic defect in OPPG.

In this study, we recruited 10 patients with OPPG and treated those who agreed (n=5) with lithium for 6 months, monitoring the response of the bones by both DXA and pQCT (peripheral quantitative computed tomography), the latter which gives information about bone quality. An IND was obtained to use lithium in this study.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria

* Age 4 years or greater
* Diagnosed with osteoporosis pseudoglioma syndrome (OPPG) or a first degree relative of someone with OPPG. For diagnosis of OPPG, one of the following is required: (1) congenital blindness in a child born into a family with known OPPG where at least one affected family member has had an LRP5 mutation demonstrated or (2) a child with no known family members with OPPG who has congenital blindness, DXA Z-score < -2.0 and mutation in LRP5 documented
* No contraindications to lithium carbonate
* For women of child bearing age, willing to undergo urine pregnancy test

Exclusion Criteria

* Age under 4 years
* Not diagnosed with osteoporosis pseudoglioma (OPPG) syndrome or a first degree relative of someone with OPPG, or a member of the Old Order Mennonite community
* Pregnant
* For women of childbearing age, not willing to undergo urine pregnancy test
* Contraindication to Lithium (serum creatinine > 1.3, known cardiovascular disease [history of myocardial infarction, heart failure], currently on diuretic or ACE inhibitor)
* Glomerular filtration rate below 80 cc/min

Ages: 4 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2010-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Streeten, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland Amish Research Clinic, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Streeten EA, McBride D, Puffenberger E, Hoffman ME, Pollin TI, Donnelly P, Sack P, Morton H. Osteoporosis-pseudoglioma syndrome: description of 9 new cases and beneficial response to bisphosphonates. Bone. 2008 Sep;43(3):584-90. doi: 10.1016/j.bone.2008.04.020. Epub 2008 May 7. PMID 18602879
- [Background] Clement-Lacroix P, Ai M, Morvan F, Roman-Roman S, Vayssiere B, Belleville C, Estrera K, Warman ML, Baron R, Rawadi G. Lrp5-independent activation of Wnt signaling by lithium chloride increases bone formation and bone mass in mice. Proc Natl Acad Sci U S A. 2005 Nov 29;102(48):17406-11. doi: 10.1073/pnas.0505259102. Epub 2005 Nov 17. PMID 16293698
- [Background] Streeten EA, Ramirez S, Eliades M, Jaimungal S, Chandrasekaran S, Kathleen R, Holmes Morton D, Puffenberger EG, Herskovitz R, Leonard MB. Fractures on bisphosphonates in osteoporosis pseudoglioma syndrome (OPPG): pQCT shows poor bone density and structure. Bone. 2015 Aug;77:17-23. doi: 10.1016/j.bone.2015.04.007. Epub 2015 Apr 16. PMID 25892485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from patients with OPPG being treated by Dr Streeten and their unaffected family members
Period: Overall Study
Arm/Group | Lithium | Unaffected Controls
Started | 10 | 16
Completed | 4 (Only 5 individuals were recruited into the Lithium treatment arm) | 16
Not Completed | 6 | 0
Not completed — 5 not started, 1 stop due to side effect | 6 | 0

BASELINE CHARACTERISTICS:
Population: All participants were from the Old Order Mennonite community from PA
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithium | Unaffected Controls | Total
Number analyzed (Participants) | 10 | 16 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 8 | 15
  Between 18 and 65 years | 3 | 8 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (2.5) | 21.8 (16.5) | 18.8 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 15
  Male | 6 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Causasian | 10 | 16 | 26
Region of Enrollment [Number; unit: participants]
  United States | 10 | 16 | 26

OUTCOME MEASURES:

1. Primary Outcome: pQCT of Lower Leg
Description: pQCT will be done at baseline for all OPPG participants and unaffecteds. The Z-score indicates the number of standard deviations away from the mean of age matched controls. A Z-score of 0 is equal to the mean, with negative numbers indicating values lower than the mean and positive values higher. A positive change in Z-score indicates a favorable outcome.
Time Frame: Baseline
Population: in OPPG, 2 were too small for pQCT machine and 2 had hardware in legs. For 2 in unaffecteds there were technical difficulties with the pQCT scanner
Measure: Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Lithium | Unaffected Controls
Number analyzed (Participants) | 10 | 16
Z-score
  Cortical Area Z-score: number analyzed (Participants) | 6 | 14
  Cortical Area Z-score | -2.19 [-3.0 to -0.14] | 0.04 [-0.51 to 0.95]
  Periosteal circum. Z | -2.09 [-3.8 to 0] | -0.30 [-2.35 to 1.17]
Statistical Analysis 1: Comparison: Lithium vs Unaffected Controls; Cortical area Z-score; Test type: Equivalence — Continuous variables were expressed as means ± SD or median (range). Group differences in pQCT Z-scores according to genotype T-test was used to compare differences at baseline between affecteds and unaffecteds; p = 0.0003, t-test, 1 sided; Differences in the two groups were assessed using Student's t-test or the rank-sum test if skewed
Statistical Analysis 2: Comparison: Lithium vs Unaffected Controls; Periosteal circumference Z-score; Test type: Equivalence — Continuous variables were expressed as means ± SD or median (range). Group differences in pQCT Z-scores according to genotype; p = 0.001, t-test, 1 sided; Differences in the two groups were assessed using Student's t-test or the rank-sum test if skewed

2. Secondary Outcome: pQCT Z-score in OPPG Participants at Baseline and 6 Months After Lithium
Description: The Z-score indicates the number of standard deviations away from the mean of age matched controls. A Z-score of 0 is equal to the mean, with negative numbers indicating values lower than the mean and positive values higher. A positive change in Z-score indicates a favorable outcome.Z-score of pQCT variable was noted for the in two OPPG participants who received lithium and were also able to get pQCT scans. The "n" of 2 was too small to do statistical analyses. Of the 5 OPPG who were on lithium, 2 were too small for the machine (eventhough over age 4) and 1 had rods in his legs and couldn't have pQCT
Time Frame: baseline, 6 months
Population: Two OPPG participants who took lithium for 6 months and were able to do pQCT at baseline and 6 months. First number is baseline, 2nd number is 6 months for section modulus
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- OPPG Rx With Lithium: Two participants who were treated with lithium and had pQCT done
Arm/Group | OPPG Rx With Lithium
Number analyzed (Participants) | 2
Z-score
  Baseline Z-score SM | -4.96 (0.12)
  6 mo Z-score SM | -4.93 (0.64)

ADVERSE EVENTS:
Time Frame: 6 months, during the administration of lithium to 5 participants
Description: Two of the participants in the lithium trial also have a severe autistic phenotype. We had hoped that the Lithium might improve their behavior. However, in one of theses 2 participants, his behavior worsened (confirmed by the Vanderbilt standardized behavioral questionnaire and he had to drop out of the study. After stopping Lithium, his behavior promptly returned to his baseline.
Arm/Group | Lithium | Unaffected Controls
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/16
Other Adverse Events (participants affected / at risk) | 1/10 | 0/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium (N=10) | Unaffected Controls (N=16)
elevated liver function test (Hepatobiliary disorders) | 1 (1) | 0 (0) — One participant who took Lithium had an elevated ALT level, present in the past prior to entry into the study and remained minimally elevated through the study. It was not felt to be related to lithium

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No